CLINICAL TRIAL: NCT06979765
Title: Research for Plasma Biomarkers Associated With Fatigue in Thrombocytopenic Patients
Acronym: FAGPLAQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: APHP240854; 2024-A01225-42 (Other: ANSM)
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Thrombopenia
Keywords: Thrombopenia
MeSH Terms: conditions — Thrombocytopenia | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): Minor patients (8 years of age or older) and adult patients seen consecutively in a hematology consultation as part of the follow-up of their thrombocytopenia.
  Interventions: Biological: blood sampling; Other: self-administrated questionaires
- Control group (Other): Control group (n=80) who will consist of healthy adult subjects (without pathology and without treatment) matched by age (± 5 years) and sex to adult patients included in the study given the possible influence of age and sex on circulating BDNF concentrations
  Interventions: Biological: blood sampling; Other: self-administrated questionaires

INTERVENTIONS:
Biological: blood sampling — 3 blood tubes will be taken during a standard check-up
Other: self-administrated questionaires — 4 self administrated questionaires and scales at the inclusion

SUMMARY:
Thrombocytopenia is a clinical problem defined by a platelet count lower than 150×10⁹/L. It can be linked to various pathologies of central origin, such as decreased platelet production in the bone marrow, or peripheral origin with increased platelet destruction through autoimmune mechanisms, increased splenic sequestration, or excessive platelet consumption. Significant fatigue is often reported in association with thrombocytopenia, but its underlying pathophysiology remains unclear. One hypothesis is the role played by neurotrophic factors contained in platelets and released into the circulation following their activation, in particular the Brain-Derived Neurotrophic Factor (BDNF), which promotes the survival, growth, differentiation, and plasticity of neurons in both the central and peripheral nervous systems. Consequently, BDNF plays a key role in long-term memory, intellectual abilities, and neuroprotection.

In this context, this project aims to confirm whether platelet-origin neurotrophic biomarkers could explain the fatigue experienced by thrombocytopenic patients and whether it depends on the etiology of the thrombocytopenia.

DETAILED DESCRIPTION:
Thrombocytopenia is defined as a platelet count below 150×109/L. The mechanisms leading to thrombocytopenia are multiple, and may be linked to :

* reduced platelet production in the bone marrow;
* increased destruction of peripheral platelets;
* increased splenic sequestration. In the event of a vascular breach, platelets contribute to hemostasis by sealing the lesion, thereby stopping bleeding. In thrombocytopenic patients, the best-known clinical signs are excessive mucocutaneous bleeding. Patients with severe thrombocytopenia (< 20×109 /L) may be at risk of life-threatening bleeding (cerebral bleeding).

In the case of autoimmune thrombocytopenia, cognitive disorders have been reported, detected by appropriate questionnaires, the pathophysiological mechanism of which remains unclear. In a study of 1871 patients with thrombocytopenia, 39% of patients in the UK and 22% in the USA reported severe asthenia. Asthenia appears to be related to thrombocytopenia, but the mechanism has not been identified either. Asthenia is a recognized symptom in other autoimmune pathologies, such as primary biliary cirrhosis (autoimmune liver disease), in which asthenia has been shown to be mainly associated with autonomic nervous system dysfunction.

While thrombocytopenia is primarily associated with bleeding risk, at least half of thrombocytopenic patients report fatigue and impaired mental and emotional health and social functioning, even though anemia is corrected and the association with autoimmune disease does not explain fatigue in all thrombocytopenic patients.

The hypothesis is that thrombocytopenia is associated with a decrease in circulating neurotrophic factor levels through reduced platelet granule secretion, which may explain the fatigue.

ELIGIBILITY:
Inclusion criteria for patients (adults or minors):

* Patients with constitutional or autoimmune (chronic or persistent ITP with last treatment administration ≥ 3 weeks) thrombocytopenia (platelet count < 150×109/L) already diagnosed
* patient not being treated and not receiving serotonin reuptake inhibitor (SSRI) or norepinephrine (SNRI) or antithrombotic treatments (antiplatelet or anticoagulant) in the 10 days prior to inclusion
* affiliation to social security (beneficiary or assignee)
* patient followed in consultation in one of the recruiting haematology departments
* Patient (or parent) having received a detailed explanation of the research project and having consent by signing the consent form before any research-specific procedure

Inclusion criteria for healthy volunteers:

* Age- (± 5 years) and sex-matched healthy adult controls
* Non-thrombocytopenic patients and not receiving antithrombotic, SNRI or SSRI therapy or if applicable, last treatment ≥ 10 days
* affiliation to social security (beneficiary or assignee)
* adults who received a detailed explanation of the research project and having consent by signing the consent form before any research-specific procedure

Non inclusion criteria (adults and minors):

* Adult patients under legal protection (guardianship or curatorship) Thrombocytopenic patients treated with antithrombotics, serotonin reuptake inhibitors (SSRIs) or noradrenaline reuptake inhibitors (SNRIs)
* Minor patients weighing less than 20 kg

Non inclusion criteria for healthy adult controls:

* Healthy adult volunteers under legal protection (guardianship, curatorship or safeguard of justice).
* Pregnant women

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2028-03-26 (Estimated); Study Completion 2028-06-26 (Estimated)

PRIMARY OUTCOMES:
Blood BDNF levels in thrombocytopenic adult and pediatric patients | At the inclusion
  Measurement of BDNF levels in thrombocytopenic patients Adults and children with excessive fatigue
Fatigue questionnaire scores for adult and pediatric patients | At the inclusion
  Fatigue questionnaire scores for adult and pediatric patients with excessive fatigue
BDNF blood level in Healthy volunteers | At the inclusion
  Measurement of BDNF blood level in Healthy volunteers

SECONDARY OUTCOMES:
Measurement of pro-BDNF blood level in thrombopenic adult and pediatric patients | At the inclusion
measurement of p75NTR blood level in thrombopenic adult and pediatric patients | At the inclusion
measurement of TrkB blood level in thrombopenic adult and pediatric patients | At the inclusion
measurement of MMP9 blood level in thrombopenic adult and pediatric patients | At the inclusion
measurement of Serotonin blood level in thrombopenic adult and pediatric patients | At the inclusion
measurement of Dopamin blood level in thrombopenic adult and pediatric patients | At the inclusion
measurement of P-selectin blood level in thrombopenic adult and pediatric patients | At the inclusion
measurement of CD40 ligand blood level in thrombopenic adult and pediatric patients | At the inclusion
anxiety questionnaire sub score of adult and pediatric patients | At the inclusion
Depression questionnaire sub score of adult and pediatric patients | At the inclusion
cognition questionnaire sub score of adult and pediatric patients | At the inclusion
measurement of pro-BDNF blood level in Healthy volunteers | At the inclusion
measurement of p75NTR blood level in Healthy volunteers | At the inclusion
measurement of TrkB blood level in Healthy volunteers | At the inclusion
measurement of MMP9 blood level in Healthy volunteers | At the inclusion
measurement of Serotonin blood level in Healthy volunteers | At the inclusion
measurement of Dopamin blood level in Healthy volunteers | At the inclusion
measurement of P-selectin blood level in Healthy volunteers | At the inclusion
measurement of CD40 ligand blood level in Healthy volunteers | At the inclusion
anxiety questionnaire sub score in Healthy volunteers | At the inclusion
Depression questionnaire sub score in Healthy volunteers | At the inclusion
cognition questionnaire sub score in Healthy volunteers | At the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Ajzenberg, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France